CLINICAL TRIAL: NCT02336893
Title: Result of an Intervention for the Group of Physicians Responsible for Providing Information on the Satisfaction of the Relatives of Patients Hospitalized in an Intensive Care Unit
Brief Title: A Semi-structured Interview PACIENTE Improves Communication With Family Members at the Intensive Care Unit
Acronym: PACIENTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DI-I-0734-13
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Communication; Quality of Life
Keywords: Communication Barriers; Total Communication Methods; Quality Improvement; Quality of Health Care; Critical Care
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-intervention (No Intervention): Family members of patients admitted to the ICU from August to December 2013 that consented to participate in the satisfaction survey and had been in the ICU for 72 h.
- Post-intervention (Experimental): Family members of patients admitted to the ICU from March to August 2014 that consented to participate in the satisfaction survey and had been in the ICU for 72 h.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — The final training was provided to a group of 34 residents --from internal medicine, anesthesiology, gynecology, and intensive care-- in charge of giving information to the patient's family members in the ICU. They were trained in the semi-structured interview PACIENTE (Present oneself and greet, Attend and listen, Call diagnosis, Inform treatment, Expose prognosis, Name introductory phrases to bad news, Take time to provide empathetic comfort, Explain an action plan involving the family) conjointly while participating in simulated difficult clinical cases with family members-actors. Four training programs were performed from February to September 2014.
  Arms: Post-intervention

SUMMARY:
The purpose of this study is to assess whether a formal training strategy using an interview PACIENTE may improve physician's skills and quality of communication with family members at the ICU.

DETAILED DESCRIPTION:
Introduction: Effective communication with physicians is an important factor for families at intensive care unit. Although physicians should have adequate communication skills, training programs are not available that would enable them to enhance this competence. Formal training using a semi-structured interview to improve skills and quality of communication was provided to physicians in charge of supplying information to families at the intensive care unit (ICU).

Objective: To assess whether a formal training strategy using an interview PACIENTE may improve physician's skills and quality of communication with family members at the ICU.

Methods: A pre- and post- intervention study was designed for a university hospital mixed ICU (medical and surgical). Training was provided to 34 resident physicians in charge of giving information to families at the ICU using interview PACIENTE. The interview was done conjointly with participation in simulated difficult clinical cases with actors posing as family members.

Patient registries: Family satisfaction was assessed with a validated survey, FS-ICU 24, in 122 and 123 family members pre- and post-intervention training, respectively, on the fourth day after patient admission to the ICU. The surveys were identified with consecutive numbers and not collected data that would allow subsequent identification of patients or their families. After the intervention, structures of interviews were monitored with checklists designed for this purpose. The meetings were always in the same place for this activity.

The surveys were answered on paper and the data included in an SPSS database by one of the researchers. Single questions in the 24-FS-ICU survey were analyzed according to the author's suggestions with minor modifications. Scores from items 1-6 in the published survey were transformed to scores from 0 to 100. The Mann-Whitney U test was used to determine any score differences between pre- and post-interventions. Differences of P<0.05 were considered statistically significant.

The sample size was calculated to be 122 participants for pre-intervention and 122 participants for post-intervention to detect α coefficient of 0.05 and with a power of 0.90. The survey was performed in the waiting room and questionnaires were collected immediately; thus, there were no missing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* That consented to participate in the satisfaction survey
* That whom had been in the ICU for 72 h.

Exclusion Criteria:

* Family members with language barriers (requiring assistance to answer a question in writing)
* Previous ICU admission within the study period
* Patient's death by the fourth day of admission
* Proved reasons for risk of judicial proceedings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Comprehension of the information, measured with the instrument FS-ICU 24. Third question, second part. | Four months
  Measured with the instrument FS-ICU 24. Third question, second part.
Adequate time to address concerns and answer questions, measured with the instrument FS-ICU 24. Tenth question, second part. | Four months
  Measured with the instrument FS-ICU 24. Tenth question, second part.

SECONDARY OUTCOMES:
Overall satisfaction with care, measured with the instrument FS-ICU 24. | Four months
  Measured with the instrument FS-ICU 24.
Overall satisfaction with decision-making measured with the instrument FS-ICU 24. | Four months
  Measured with the instrument FS-ICU 24.
Global survey satisfaction measured with the instrument FS-ICU 24. | Four months
  Measured with the instrument FS-ICU 24.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel H Coral, MD, Principal Investigator — Fundación Universitaria de Ciencias de la Salud

REFERENCES:
- [Result] Fumis RR, Nishimoto IN, Deheinzelin D. Families' interactions with physicians in the intensive care unit: the impact on family's satisfaction. J Crit Care. 2008 Sep;23(3):281-6. doi: 10.1016/j.jcrc.2007.04.004. Epub 2007 Jul 5. PMID 18725030
- [Result] Bailey JJ, Sabbagh M, Loiselle CG, Boileau J, McVey L. Supporting families in the ICU: a descriptive correlational study of informational support, anxiety, and satisfaction with care. Intensive Crit Care Nurs. 2010 Apr;26(2):114-22. doi: 10.1016/j.iccn.2009.12.006. Epub 2010 Jan 27. PMID 20106664
- [Result] Karlsson C, Tisell A, Engstrom A, Andershed B. Family members' satisfaction with critical care: a pilot study. Nurs Crit Care. 2011 Jan-Feb;16(1):11-8. doi: 10.1111/j.1478-5153.2010.00388.x. PMID 21199550
- [Result] Curtis JR, Engelberg RA, Wenrich MD, Nielsen EL, Shannon SE, Treece PD, Tonelli MR, Patrick DL, Robins LS, McGrath BB, Rubenfeld GD. Studying communication about end-of-life care during the ICU family conference: development of a framework. J Crit Care. 2002 Sep;17(3):147-60. doi: 10.1053/jcrc.2002.35929. PMID 12297990
- [Result] Azoulay E, Pochard F, Chevret S, Lemaire F, Mokhtari M, Le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Meeting the needs of intensive care unit patient families: a multicenter study. Am J Respir Crit Care Med. 2001 Jan;163(1):135-9. doi: 10.1164/ajrccm.163.1.2005117. PMID 11208638
- [Result] Brown A, Hijazi M. Arabic translation and adaptation of Critical Care Family Satisfaction Survey. Int J Qual Health Care. 2008 Aug;20(4):291-6. doi: 10.1093/intqhc/mzn013. Epub 2008 Apr 10. PMID 18403569
- [Result] Auerbach SM, Kiesler DJ, Wartella J, Rausch S, Ward KR, Ivatury R. Optimism, satisfaction with needs met, interpersonal perceptions of the healthcare team, and emotional distress in patients' family members during critical care hospitalization. Am J Crit Care. 2005 May;14(3):202-10. PMID 15840894
- [Result] Alexander SC, Keitz SA, Sloane R, Tulsky JA. A controlled trial of a short course to improve residents' communication with patients at the end of life. Acad Med. 2006 Nov;81(11):1008-12. doi: 10.1097/01.ACM.0000242580.83851.ad. PMID 17065871
- [Result] Lorin S, Rho L, Wisnivesky JP, Nierman DM. Improving medical student intensive care unit communication skills: a novel educational initiative using standardized family members. Crit Care Med. 2006 Sep;34(9):2386-91. doi: 10.1097/01.CCM.0000230239.04781.BD. PMID 16791111
- [Result] Back AL, Arnold RM, Baile WF, Fryer-Edwards KA, Alexander SC, Barley GE, Gooley TA, Tulsky JA. Efficacy of communication skills training for giving bad news and discussing transitions to palliative care. Arch Intern Med. 2007 Mar 12;167(5):453-60. doi: 10.1001/archinte.167.5.453. PMID 17353492
- [Result] Sullivan AM, Lakoma MD, Billings JA, Peters AS, Block SD; PCEP Core Faculty. Teaching and learning end-of-life care: evaluation of a faculty development program in palliative care. Acad Med. 2005 Jul;80(7):657-68. doi: 10.1097/00001888-200507000-00008. PMID 15980082
- [Result] Fineberg IC. Preparing professionals for family conferences in palliative care: evaluation results of an interdisciplinary approach. J Palliat Med. 2005 Aug;8(4):857-66. doi: 10.1089/jpm.2005.8.857. PMID 16128661
- [Result] Shaw DJ, Davidson JE, Smilde RI, Sondoozi T, Agan D. Multidisciplinary team training to enhance family communication in the ICU. Crit Care Med. 2014 Feb;42(2):265-71. doi: 10.1097/CCM.0b013e3182a26ea5. PMID 24105452
- [Result] Baile WF, Buckman R, Lenzi R, Glober G, Beale EA, Kudelka AP. SPIKES-A six-step protocol for delivering bad news: application to the patient with cancer. Oncologist. 2000;5(4):302-11. doi: 10.1634/theoncologist.5-4-302. PMID 10964998
- [Result] Azoulay E, Pochard F, Chevret S, Arich C, Brivet F, Brun F, Charles PE, Desmettre T, Dubois D, Galliot R, Garrouste-Orgeas M, Goldgran-Toledano D, Herbecq P, Joly LM, Jourdain M, Kaidomar M, Lepape A, Letellier N, Marie O, Page B, Parrot A, Rodie-Talbere PA, Sermet A, Tenaillon A, Thuong M, Tulasne P, Le Gall JR, Schlemmer B; French Famirea Group. Family participation in care to the critically ill: opinions of families and staff. Intensive Care Med. 2003 Sep;29(9):1498-504. doi: 10.1007/s00134-003-1904-y. Epub 2003 Jul 10. PMID 12856124
- [Result] Wall RJ, Engelberg RA, Downey L, Heyland DK, Curtis JR. Refinement, scoring, and validation of the Family Satisfaction in the Intensive Care Unit (FS-ICU) survey. Crit Care Med. 2007 Jan;35(1):271-9. doi: 10.1097/01.CCM.0000251122.15053.50. PMID 17133189
- [Result] Heyland DK, Tranmer JE; Kingston General Hospital ICU Research Working Group. Measuring family satisfaction with care in the intensive care unit: the development of a questionnaire and preliminary results. J Crit Care. 2001 Dec;16(4):142-9. doi: 10.1053/jcrc.2001.30163. PMID 11815899